CLINICAL TRIAL: NCT04289675
Title: Chi3L1: A Marker of Efficacy of Platform Treatments in Relapsing-onset Multiple Sclerosis: A Prognostic Study on Existing Clinical Data and Biological Samples
Brief Title: Multiple Sclerosis: Chi3L1 and Treatment Efficacy
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: CPRC 2018 / CHI3L1-MATHEY/MS
Record Dates: First submitted 2019-12-27; First posted 2020-02-28 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2019-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon-beta; Dimethyl Fumarate; teriflunomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Blood samples : chitinase 3-like 1 level Cerebrospinal fluid samples : chitinase 3-like 1, neurofilaments light chains and interleukin 6 levels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Interferon-Beta: Patients with first treatment : interferon beta (1a subcutaneous 22 or 44 µg thrice a week OR 1a intramuscular 30 µg once a week OR 1b subcutaneous 250 µg every other day OR 1a PEGylated subcutaneous 125 µg every two weeks)
  Interventions: Drug: Interferon-Beta
- Dimethyl fumarate: Patients with first treatment : dimethyl fumarate (oral, 240 mg twice a day)
- Teriflunomide: Patients with first treatment : teriflunomide (oral, 14 mg once a day)

INTERVENTIONS:
Drug: Interferon-Beta — Theses drugs have been administered as part of routine care. Biological samples that will be analyzed (blood and cerebrospinal fluid) have been taken as part of routine care.
  Other Names: Dimethyl fumarate; Teriflunomide
  Groups: Interferon-Beta

SUMMARY:
Chitinase 3-like 1 (Chi3L1) is a Human protein synthetized by inflammatory cells. Its serum level increases in case of autoimmune diseases, and especially during multiple sclerosis (MS). There is a need for biological markers predictive of treatment efficacy. MS outcomes one year from treatment initiation are predictive of long-term treatment efficacy. The hypothesis is that serum Chi3L1 level before treatment initiation could predict one year MS outcomes.

Primary objective: to show an association between the serum Chi3L1 level at diagnostic assessment and the clinical and radiological efficacy one year from initiation of the first disease modifying treatment (interferon beta, dimethyl fumarate or teriflunomide) in relapsing-onset multiple sclerosis (MS).

Secondary objectives: to determine the threshold value of the serum Chi3L1 level predicting the efficacy of treatment, and the added value of other potential biomarkers in cerebrospinal fluid collected at diagnostic assessment: Chi3L1, light chains of neurofilaments and interleukin 6.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-onset multiple sclerosis according to the 2017 McDonald criteria
* Blood and cerebrospinal fluid samples collected at diagnostic assessment from 2012 January 1st and kept in the Centre de Ressources Biologiques Lorrain
* First platform disease modifying drugs : interferon-Beta, dimethyl fumarate or teriflunomide, introduced during the first 3 months after the diagnostic assessment
* Disease modifying drugs maintained at least 3 months
* Follow-up during at least 15 months after the first disease modifying drug initiation
* At least one brain magnetic resonance imaging with gadolinium injection between months 3 and 15 after disease modifying drug initiation

Exclusion Criteria:

* Objection to the use of personal data for research purpose

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Patients are selected from the Registre Lorrain des Scléroses en Plaques (ReLSEP). Demographical, clinical and paraclinical data are already collected in this database. Biological tests will be performed on their relative blood and cerebrospinal fluid samples, already taken and kept in the Centre de Ressources Biologiques Lorrain.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Statistical association between the baseline chitinase 3-like 1 serum level and being "responder" at year one | Baseline to month 15
  Significant associations in each group of treatment
  Being "responder" means the presence of the four following :
  * No treatment withdrawal between months 3 and 15 after treatment initiation for reason of inefficacy
  * No relapse between months 3 and 15
  * No increase of at least one point on the expanded disability status scale between months 3 and 15
  * No gad-enhancing lesion on any magnetic resonance imaging scan between months 3 and 15
  If any of these criteria is lacking, then the patient is considered as "non-responder".

SECONDARY OUTCOMES:
Threshold chitinase 3-like 1 serum level at baseline to distinguish responders from non-responders | Baseline to month 15
  Threshold measure that discriminates responders and non-responders at month 15 in each group
Statistical association between the baseline chitinase 3-like 1 cerebrospinal fluid level and being "responder" at year one | Baseline to month 15
  Significant associations in each group of treatment
  Being "responder" means the presence of the four following :
  * No treatment withdrawal between months 3 and 15 after treatment initiation for reason of inefficacy
  * No relapse between months 3 and 15
  * No increase of at least one point on the expanded disability status scale between months 3 and 15
  * No gad-enhancing lesion on any magnetic resonance imaging scan between months 3 and 15
  If any of these criteria is lacking, then the patient is considered as "non-responder".
Statistical association between the baseline neurofilaments light chains cerebrospinal fluid level and being "responder" at year one | Baseline to month 15
  Significant associations in each group of treatment
  Being "responder" means the presence of the four following :
  * No treatment withdrawal between months 3 and 15 after treatment initiation for reason of inefficacy
  * No relapse between months 3 and 15
  * No increase of at least one point on the expanded disability status scale between months 3 and 15
  * No gad-enhancing lesion on any magnetic resonance imaging scan between months 3 and 15
  If any of these criteria is lacking, then the patient is considered as "non-responder".
Statistical association between the baseline interleukin 6 cerebrospinal fluid level and being "responder" at year one | Baseline to month 15
  Significant associations in each group of treatment
  Being "responder" means the presence of the four following :
  * No treatment withdrawal between months 3 and 15 after treatment initiation for reason of inefficacy
  * No relapse between months 3 and 15
  * No increase of at least one point on the expanded disability status scale between months 3 and 15
  * No gad-enhancing lesion on any magnetic resonance imaging scan between months 3 and 15
  If any of these criteria is lacking, then the patient is considered as "non-responder".

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Mathey, MSc, MD, Principal Investigator — Hôpital Central - service de Neurologie - CHRU Nancy

IPD SHARING:
Plan to Share IPD: No